CLINICAL TRIAL: NCT02458885
Title: Relevamiento / Encuesta Nacional de Infarto Agudo de Miocardio Con elevación Del ST
Brief Title: Pilot Study on ST Elevation Acute Myocardial Infarction
Acronym: ARGEN-IAM-ST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sociedad Argentina de Cardiología (Other)
Collaborators: Federación Argentina de Cardiología (Unknown)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2015-05-26; First posted 2015-06-01 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; observational registry; mortality
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aim of investigators is to conduct a registry of acute myocardial infarction including a broad network of critical care / coronary care unit throughout Argentina to increase the knowledge about treatments, timing of reperfusion therapy and outcomes, both in-hospital and during short-term follow up.

DETAILED DESCRIPTION:
Cardiovascular disease is the most common cause of death in the world and in Argentina, as well as a cause of disability and loss of work capacity in adults. Treatment of various forms of serious diseases such as acute ischemic events and heart failure are now supported by scientific studies and allow a markedly reduction in disability and mortality. Access to diagnostic and therapeutic strategies require proper coordination of the health system and far exceed the role of specialists. Given the frequency of these diseases, it is essential to have information on the prevalence and treatment, and the various barriers to access to diagnosis and appropriate treatment. Both for the basic knowledge to evaluate the relevance and effectiveness of corrective action a record of pathologies is required, with information accurate enough to enable the adoption of public policies, and adjusted to national needs.

Scientific societies in cardiovascular field, Argentine Society of Cardiology and Argentine Federation of Cardiology, have a long history of registers and educational programs to improve cardiovascular care. However, these tasks are limited to institutions with academic programs and probably do not reach the majority of our population.

A national survey of high prevalence of cardiovascular diseases, starting with acute myocardial infarction with ST segment elevation, together with the authorities of the National Ministry of Health, would put Argentina at the level of most developed countries in this subject. Knowledge of general and local barriers will allow a rapid implementation of corrective measures and the evaluation of their impact through the permanent record. Improving the quality of cardiovascular patient care, optimizing adherence to standards of diagnosis and treatment can be achieved through different paths as self-knowledge of the institutions of their level of performance and dissemination of coordination measures, generating systematic referral and care networks, diagnostic support systems such as telemedicine, and others that can be assessed globally or regionally according to the identified problems.

Networking will also enable the implementation of initiatives that will result in an increase in the quality of care and generate epidemiological research projects that enhance patient care and outcomes. In conclusion, it will allow to know the problems in depth and adopt measures to improve the quality of care and reduce morbidity and mortality.

The main objective of the survey is to register at national level, in the broadest possible way trying to reach the "universe" of care for this disease in Argentina, aspects of clinical, delays, treatment schedules and results, with sufficient information to quickly allow the adoption of policies to improve the quality of care and subsequent control.

Its fulfilment arises in stages:

1. Develop a national survey of myocardial infarction with ST segment elevation, aimed at characterization of current evolutions and possible barriers to be improved.
2. Based on the results, configure an advisory group for public policies in this area to suggest global and regional measures.
3. Upon completion of the survey, consolidation of a permanent network of cardiovascular disease registry to assess the impact of public policies and their progressive adjustment under the Federal Cardiovascular Disease Registry A national survey of all AMI with ST segment elevation admitted to intensive care areas across the country will take place over a period of 3 consecutive months in each centre.

The inclusion criteria are:

* Patients admitted with AMI and ST-segment elevation.
* AMI evolved with new Q waves less than 36 hours evolution.
* Suspected inferoposterior AMI (horizontal ST depression in V1 to V3, suggestive of acute circumflex coronary artery occlusion).
* New or presumed new left bundle branch block.

Exclusion criteria:

* Acute coronary syndrome without ST elevation or non-Q AMI
* Myocardial infarction of more than 36 hours of evolution. Data on patient characteristics (age, gender, risk factors, history, comorbidities), of the clinical conditions (infarct location, Killip on admission, duration of symptoms), treatments (antiplatelet drugs, reperfusion therapy, adjuvant treatment) and in-hospital (heart failure, post-infarction angina, shock, death) and 30-day evolution will be collected. Emphasis will be placed on the delays for effective treatment. 30 days follow-up will be done by telephone or in person by each centre investigator or through the central coordinating committee.

The data collection will take place in an electronic record specially designed, via web, allowing constant monitoring of the input data. The survey data will be verified or confronted with source documents in at least 30% of the patients included in the survey.

The data analysis will be conducted by a committee of representatives of the organizing researchers of Scientific Societies and the Ministry of Health, presented in relevant scientific meetings and published in the journals of both Societies.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with AMI and ST-segment elevation.
* AMI evolved with new Q waves less than 36 hours evolution.
* Suspected inferoposterior AMI (horizontal ST depression in V1 to V3, suggestive of acute circumflex coronary artery occlusion).
* New or presumed new left bundle branch block.

Exclusion Criteria:

* Acute coronary syndrome without ST elevation or non-Q AMI
* Myocardial infarction of more than 36 hours of evolution.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ST elevation Myocardial infarction.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Appropriate use of reperfusion therapy | In-hospital, with an expected average of 5 days.
  Timely initiation of reperfusión (door to needle time <30 minutes or door to balloon time <90 minutes).
In-hospital mortality | In-hospital, with an expected average of 5 days.
  All cause death during initial hospitalization.
All cause mortality | 30 days.
  All cause mortality between symptoms onset and 30 days.

SECONDARY OUTCOMES:
In-hospital complications | In-hospital, with an expected average of 5 days.
  Heart failure, post-infarction angina, cardiogenic shock or death during initial hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gagliardi, PhD, Study Chair — +54 114961-6027
Locations (1):
- Sociedad Argentina de Cardiología, Ciudad Autónoma de Buenos Aires, Buenos Aires, Argentina